CLINICAL TRIAL: NCT02378103
Title: A Single-center Trial of Patients With Aortic Dissection in the Chinese XinJiang Province
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Xiang Ma (Other)
Responsible Party: Sponsor-Investigator, Xiang Ma, A Single-center Trial of Patients with Aortic Dissection in the Chinese XinJiang Province, First Affiliated Hospital of Xinjiang Medical University
Organization: First Affiliated Hospital of Xinjiang Medical University (Other)
Other Study IDs: IACUC-20140214090
Record Dates: First submitted 2015-02-14; First posted 2015-03-04 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Aortic Dissection
Keywords: Aortic Dissection; Chinese XinJiang Province
MeSH Terms: conditions — Aortic Dissection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Case: Diagnosis of aortic dissection was based on history and physical examination, and confirmed by imaging, visualization at surgery, and/or postmortem examination. Simple aortic aneurysm and pseudoaneurysm were excluded. Simple aortic aneurysm and pseudoaneurysm were excluded. Surgical and endovascular treatments were the main interventions and performed in the case group.
- Control: As the control group, patients without AD were obtained from the hospitalized patients in the same period.

SUMMARY:
To evaluate epidemiological features of risk factors for aortic dissection (AD) in Chinese XinJiang Province patients.

DETAILED DESCRIPTION:
The epidemiological features of risk factors for aortic dissection (AD) in China were obtained from developed population in east of China, however, such information was not available for the remote population. Moreover, people in the western region have significant difference with developed population in lifestyle, diet, ethnic and so on. Therefore, the aim of our study was to evaluate epidemiological features of risk factors for AD in Chinese remote patients. We anticipated that this analysis would provide helpful information preventing and controlling AD in Chinese XinJiang Province.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of aortic dissection
2. ≥18 years old
3. good compliance with the instructions and cooperate with follow-up voluntarily signed the informed consent form

Exclusion Criteria:

1. pregnant or lactating female
2. bad compliance with the instructions and follow-up
3. estimated remaining life is less than 12 months
4. Aortic aneurysm、Acute Myocardial infarction、Acute Cerebral accident

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Between March, 2015 and March, 2016, we aim to collect 100 patients with AD as the case group. As the control group, 100 patients without AD were obtained from the hospitalized patients in the same period.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-02; Primary Completion 2016-03 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Participants with related events for aortic dissection in Chinese XinJiang population | 1 year